CLINICAL TRIAL: NCT01189604
Title: A Multi-centre, Single-blind, Randomised, Parallel Group, Phase IIb Dose Rate Range Finding Study to Find Maintenance Dose Rate Range of ICI35,868 for the Minimal-to-moderate Sedation on Gastrointestinal Endoscopic Tests (Including Endoscopic Polypectomy)
Brief Title: Dose Rate Range Finding Study of Propofol for minimal-to Moderate Sedation on Upper & Lower Endoscopic Tests
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Johnson & Johnson K.K. Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D0092C00001
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Gastrointestinal Endoscopy; Gastrointestinal Polypectomy
Keywords: propofol endoscopy sedation
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (7):
- Arm1 - Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 2 - ICI35,868 (propofol) (Active Comparator)
  Interventions: Drug: ICI35,868 (propofol)
- Arm 3 - ICI35,868 (propofol) (Active Comparator)
  Interventions: Drug: ICI35,868 (propofol)
- Arm 4 - ICI35,868 (propofol) (Active Comparator)
  Interventions: Drug: ICI35,868 (propofol)
- Arm 5 - ICI35,868 (propofol) (Active Comparator)
  Interventions: Drug: ICI35,868 (propofol)
- Arm 6 - ICI35,868 (propofol) (Active Comparator)
  Interventions: Drug: ICI35,868 (propofol)
- Arm 7 - ICI35,868 (propofol) (Active Comparator)
  Interventions: Drug: ICI35,868 (propofol)

INTERVENTIONS:
Drug: Placebo — Infusion of placebo, same infusion rates as for arm 2
  Arms: Arm1 - Placebo
Drug: ICI35,868 (propofol) — Infusion of propofol: initiation with 0.17 mg/kg for 3 minutes followed by maintenance with 25 µg/kg/minute
  Arms: Arm 2 - ICI35,868 (propofol)
Drug: ICI35,868 (propofol) — Infusion of propofol: initiation with 0.33 mg/kg for 3 minutes followed by maintenance with 50 µg/kg/minute
  Arms: Arm 3 - ICI35,868 (propofol)
Drug: ICI35,868 (propofol) — Infusion of propofol: initiation with 0.5 mg/kg for 3 minutes followed by maintenance with 75 µg/kg/minute
  Arms: Arm 4 - ICI35,868 (propofol)
Drug: ICI35,868 (propofol) — Infusion of propofol: initiation with 0.8 mg/kg for 3 minutes followed by maintenance with 120 µg/kg/minute
  Arms: Arm 5 - ICI35,868 (propofol)
Drug: ICI35,868 (propofol) — Infusion of propofol: initiation with 0.5 mg/kg for 1 minutes followed by maintenance with 75 µg/kg/minute
  Arms: Arm 6 - ICI35,868 (propofol)
Drug: ICI35,868 (propofol) — Infusion of propofol: initiation with 0.5 mg/kg for 5 minutes followed by maintenance with 75 µg/kg/minute
  Arms: Arm 7 - ICI35,868 (propofol)

SUMMARY:
Phase IIB study to find the optimal dose rate range of propofol to maintain minimal-to-moderate sedation for diagnostic gastrointestinal endoscopy and gastrointestinal polypectomy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female (females of child bearing potential to confirm not pregnant via test or contraception)
* Be undergoing a non-emergent esophagogastroduodenoscopy (EGD) or colonoscopy, including polypectomy that shall be completed within 1 hour

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) grade III, IV V and VI
* Baseline oxygen saturation<90% (room air)
* Body Mass Index (BMI) >=35

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2010-08; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masataka Date, M.D., Ph.D., Study Director — Physician Group, Clinical Division, R&D, Astrazeneca K.K.
Locations (2):
- Japan (2):
  - Research Site, Isesaki, Gunma
  - Research Site, Moriya, Ibaragi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 2 centers were initiated with first patient enrolled on 23 August 2010 and last patient completed on 17 November. A total of 129 patients were enrolled with 123 qualified patients allocated to randomized treatment.
Pre-assignment Details: The patients enrolled in this study were undergoing non-emergent standard esophagogastroduodenoscopy (EGD) or colonoscopy. Six patients were withdrawn from the study after enrollment but before randomization: 5 patients due to excess recruitment and one patient due to investigator's recommendation..
Groups:
- Arm 1 - Placebo: Infusion of placebo, same infusion rates as for arm 2
- Arm 2 - ICI35,868 (Propofol): Infusion of propofol: initiation with 0.17 mg/kg for 3 minutes followed by maintenance with 25 µg/kg/minute
- Arm 3 - ICI35,868 (Propofol): Infusion of propofol: initiation with 0.33 mg/kg for 3 minutes followed by maintenance with 50 µg/kg/minute
- Arm 4 - ICI35,868 (Propofol): Infusion of propofol: initiation with 0.5 mg/kg for 3 minutes followed by maintenance with 75 µg/kg/minute
- Arm 5 - ICI35,868 (Propofol): Infusion of propofol: initiation with 0.8 mg/kg for 3 minutes followed by maintenance with 120 µg/kg/minute
- Arm 6 - ICI35,868 (Propofol): Infusion of propofol: initiation with 0.5 mg/kg for 1 minutes followed by maintenance with 75 µg/kg/minute
- Arm 7 - ICI35,868 (Propofol): Infusion of propofol: initiation with 0.5 mg/kg for 5 minutes followed by maintenance with 75 µg/kg/minute
Period: Overall Study
Arm/Group | Arm 1 - Placebo | Arm 2 - ICI35,868 (Propofol) | Arm 3 - ICI35,868 (Propofol) | Arm 4 - ICI35,868 (Propofol) | Arm 5 - ICI35,868 (Propofol) | Arm 6 - ICI35,868 (Propofol) | Arm 7 - ICI35,868 (Propofol)
Started | 21 | 21 | 20 | 20 | 20 | 11 | 10
Administered Study Drug | 20 | 20 | 20 | 20 | 20 | 10 | 10
Completed | 20 | 20 | 20 | 20 | 18 | 10 | 9
Not Completed | 1 | 1 | 0 | 0 | 2 | 1 | 1
Not completed — Impossible to visit | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 - Placebo | Arm 2 - ICI35,868 (Propofol) | Arm 3 - ICI35,868 (Propofol) | Arm 4 - ICI35,868 (Propofol) | Arm 5 - ICI35,868 (Propofol) | Arm 6 - ICI35,868 (Propofol) | Arm 7 - ICI35,868 (Propofol) | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 10 | 10 | 120
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (17.3) | 51.0 (16.4) | 56.1 (14.4) | 52.0 (14.9) | 56.4 (12.7) | 49.4 (14.2) | 51.8 (8.5) | 53.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 10 | 6 | 9 | 2 | 5 | 48
  Male | 14 | 10 | 10 | 14 | 11 | 8 | 5 | 72
Procedures [Number; unit: participants] — Patients underwent either esophagogastroduodenoscopy (EGD) or colonoscopy.
  participants
    Esophagogastroduodenoscopy (EGD) | 10 | 10 | 10 | 10 | 10 | 5 | 5 | 60
    Colonoscopy | 10 | 10 | 10 | 10 | 10 | 5 | 5 | 60

OUTCOME MEASURES:

1. Primary Outcome: Modified Observers Assessment of Alertness/Sedation (MOAA/S) Score 2 Minutes From Beginning of Maintenance Period
Description: The MOAA/S is a 6-point ordinal scale measuring a patient's level of sedation. Scores range from 0 (No response to painful stimulus [trapezius squeeze]) to 5 (Responds readily to name spoken in normal tone [awake]). MOAA/S scores were classified as 0-1, 2-4 and 5.
Time Frame: 2 minutes from the beginning of the maintenance period
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - ICI35,868 (Propofol) | Arm 3 - ICI35,868 (Propofol) | Arm 4 - ICI35,868 (Propofol) | Arm 5 - ICI35,868 (Propofol) | Arm 6 - ICI35,868 (Propofol) | Arm 7 - ICI35,868 (Propofol)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 10 | 10
Participants
  MOAA/S Score 0-1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  MOAA/S Score 2-4 | 0 | 2 | 6 | 6 | 14 | 5 | 3
  MOAA/S Score 5 | 20 | 18 | 14 | 13 | 5 | 4 | 7

2. Primary Outcome: Modified Observers Assessment of Alertness/Sedation (MOAA/S) Score 4 Minutes From Beginning of Maintenance Period
Description: as for outcome 1
Time Frame: 4 minutes from the beginning of the maintenance period
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - ICI35,868 (Propofol) | Arm 3 - ICI35,868 (Propofol) | Arm 4 - ICI35,868 (Propofol) | Arm 5 - ICI35,868 (Propofol) | Arm 6 - ICI35,868 (Propofol) | Arm 7 - ICI35,868 (Propofol)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 10 | 10
Participants
  MOAA/S Score 0-1 | 0 | 0 | 0 | 1 | 3 | 1 | 0
  MOAA/S Score 2-4 | 0 | 1 | 7 | 6 | 16 | 5 | 4
  MOAA/S Score 5 | 20 | 19 | 13 | 13 | 1 | 4 | 6

3. Secondary Outcome: Patient Satisfaction With Sedation Instrument (PSSI) Questionnaire
Description: The PSSI is a 100-point visual analog scale measuring a patient's satisfaction with sedation. Scores range from 0 (Very dissatisfied) to 100 (Very satisfied).
Time Frame: 24 - 48 hours after completion of the procedure
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Arm 1 - Placebo | Arm 2 - ICI35,868 (Propofol) | Arm 3 - ICI35,868 (Propofol) | Arm 4 - ICI35,868 (Propofol) | Arm 5 - ICI35,868 (Propofol) | Arm 6 - ICI35,868 (Propofol) | Arm 7 - ICI35,868 (Propofol)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 10 | 10
Units on a scale | 62.5 (21.2) | 64.4 (23.8) | 74.5 (17.1) | 82.3 (17.9) | 86.0 (9.8) | 74.9 (16.2) | 75.1 (21.2)

4. Secondary Outcome: Blood Concentrations of Propofol
Description: Blood concentration of ICI35,868 (propofol)
Time Frame: At the end of the initiation period and every 2 minutes during the maintenance period
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Arm 1 - Placebo | Arm 2 - ICI35,868 (Propofol) | Arm 3 - ICI35,868 (Propofol) | Arm 4 - ICI35,868 (Propofol) | Arm 5 - ICI35,868 (Propofol) | Arm 6 - ICI35,868 (Propofol) | Arm 7 - ICI35,868 (Propofol)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 4 | 4
µg/mL
  End of initiation period |  | 0.2208 (0.1409) | 0.7808 (0.3765) | 1.5033 (0.9468) | 2.3177 (1.2459) | 1.1935 (1.0758) | 1.0875 (0.7553)
  2 minutes into maintenance period |  | 0.2797 (0.1320) | 0.6403 (0.3087) | 1.1052 (0.7197) | 2.1827 (0.7832) | 1.3965 (0.7796) | 0.8515 (0.6399)
  4 minutes into maintenance period |  | 0.3295 (0.1474) | 0.7387 (0.3000) | 1.2022 (0.5612) | 2.4360 (0.8500) | 1.4828 (0.4286) | 1.0708 (0.7864)
  6 minutes into maintenance period |  | 0.3633 (0.2340) | 0.8127 (0.2716) | 1.4263 (0.6700) | 2.4714 (0.3901) | 1.4848 (0.4056) | 1.0560 (0.7915)

5. Secondary Outcome: Modified Observers Assessment of Alertness/Sedation (MOAA/S) at End of Initiation Period
Description: as for outcome 1
Time Frame: Last measurement in maintenance period (3 minutes for arms 1-5; 1 minute for arm 6, 5 minute for arm 7)
Measure: Number; unit: Participants
Arm/Group | Arm 1 - Placebo | Arm 2 - ICI35,868 (Propofol) | Arm 3 - ICI35,868 (Propofol) | Arm 4 - ICI35,868 (Propofol) | Arm 5 - ICI35,868 (Propofol) | Arm 6 - ICI35,868 (Propofol) | Arm 7 - ICI35,868 (Propofol)
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 10 | 10
Participants
  MOAA/S Score 0-1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  MOAA/S Score 2-4 | 0 | 2 | 0 | 4 | 9 | 0 | 1
  MOAA/S Score 5 | 20 | 18 | 20 | 16 | 10 | 10 | 9

ADVERSE EVENTS:
Arm/Group | Arm 1 - Placebo | Arm 2 - ICI35,868 (Propofol) | Arm 3 - ICI35,868 (Propofol) | Arm 4 - ICI35,868 (Propofol) | Arm 5 - ICI35,868 (Propofol) | Arm 6 - ICI35,868 (Propofol) | Arm 7 - ICI35,868 (Propofol)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 5/20 | 0/20 | 0/20 | 1/20 | 6/20 | 1/10 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 - Placebo (N=20) | Arm 2 - ICI35,868 (Propofol) (N=20) | Arm 3 - ICI35,868 (Propofol) (N=20) | Arm 4 - ICI35,868 (Propofol) (N=20) | Arm 5 - ICI35,868 (Propofol) (N=20) | Arm 6 - ICI35,868 (Propofol) (N=10) | Arm 7 - ICI35,868 (Propofol) (N=10)
Ventricular Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood Pressure Decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood Pressure Increased (Investigations) | 4 | 0 | 0 | 0 | 0 | 0 | 0
C-Reactive Protein Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart Rate Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Angiopathy (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the PI wants to publish the results, the PI must send the English documents to AZ beforehand. And AZ can review and revise the documents, after that, AZ will give the approval to the PI about the publication of the results.